CLINICAL TRIAL: NCT01757054
Title: Randomized, Two Arm, Parallel Group, Open Label, Single Center Prospective Study of the Fecal Recovery of Lactobacillus Rhamnosus GG (LGG) and Bifidobacterium Animalis Subspecies Lactis (BB-12) in Healthy Humans Following Daily Consumption of ProNutrients Probiotic Powder Sachet
Brief Title: Fecal Recovery of the Probiotic Bacteria Lactobacillus Rhamnosus GG (LGG) and Bifidobacterium Animalis Subspecies Lactis BB-12 (BB-12) in Healthy Humans Following Daily Consumption of a Probiotic Supplement
Acronym: LGG BB-12
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: B4141001; PO-10-08
Record Dates: First submitted 2012-12-20; First posted 2012-12-28 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Fecal Analysis
Keywords: probiotic; LGG; BB-12; fecal recovery; healthy subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic group (Experimental)
  Interventions: Dietary Supplement: ProNutrients Probiotic
- Control group (No Intervention): This is a non-supplemented control group that will follow the same dietary and medication restrictions. The purpose of this group is to ensure results are due to supplementation and not due to random dietary exposure.

INTERVENTIONS:
Dietary Supplement: ProNutrients Probiotic — Dosage is 1 individually wrapped packet (1 gram) containing probiotic powder per day for 21 days
  Arms: Probiotic group

SUMMARY:
The main hypothesis of this study is that there will be a significant increase of Lactobacillus rhamnosus GG (LGG) and Bifidobacterium lactis (BB-12) in the stool of healthy humans following daily consumption of a probiotic supplement containing these specific strains of probiotic bacteria.

DETAILED DESCRIPTION:
To demonstrate recovery of live probiotic bacteria in the stool.

ELIGIBILITY:
Inclusion Criteria:

Are between 18-70 years of age. Have regular bowel movements. Are willing and able to attend study visits, undergo limited blood and urine testing, take the nutritional supplement according to the instructions provided.

Are willing to collect four stool specimens and bring them to the study site.

Exclusion Criteria:

Are unwilling to follow the dietary guidelines of the study. Are lactose-intolerant or have allergies to milk or wheat. Have had drug or alcohol problems within the previous year. Are or plan to become pregnant over the next 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in fecal concentration of both LGG and BB-12 by quantitative culture with confirmatory PCR at baseline and 3 weeks | Baseline, 3 weeks
  Pre- to post-supplementation changes in fecal concentration of both LGG and BB-12 by quantitative culture with confirmatory PCR

SECONDARY OUTCOMES:
Change in fecal concentration of both LGG and BB-12 by quantitative culture with confirmatory PCR at baseline and 2 weeks | Baseline, 2 weeks
  Pre- to post-supplementation changes in fecal concentration of both LGG and BB-12 by quantitative culture with confirmatory PCR
Change in fecal concentration of both LGG and BB-12 by quantitative PCR (qPCR) at baseline and 3 weeks | Baseline, 3 weeks
  Pre- to post-supplementation changes in fecal concentration of both LGG and BB-12 by quantitative PCR (qPCR)
Change in fecal concentration of both LGG and BB-12 by quantitative PCR (qPCR) at baseline and 2 weeks | Baseline, 2 weeks
  Pre- to post-supplementation changes in fecal concentration of both LGG and BB-12 by quantitative PCR (qPCR)
Change in fecal concentration of both LGG and BB-12 by quantitative culture with confirmatory PCR and qPCR in probiotic compared to control group at baseline and 3 weeks | Baseline, 3 weeks
  Pre- to post-supplementation changes in fecal concentration of both LGG and BB-12 by quantitative culture with confirmatory PCR and qPCR in probiotic compared to control group
Change in fecal concentration of both LGG and BB-12 by quantitative culture with confirmatory PCR and qPCR in probiotic compared to control group at baseline and 2 weeks | Baseline, 2 weeks
  Pre- to post-supplementation changes in fecal concentration of both LGG and BB-12 by quantitative culture with confirmatory PCR and qPCR in probiotic compared to control group
Change in fecal concentration of LGG and BB-12 by both quantitative culture with confirmatory PCR and qPCR at baseline, 3 weeks, and 28 days post supplementation | Baseline, 3 weeks, 28 days follow up
  Post-supplementation fecal concentration of LGG and BB-12 by both quantitative culture with confirmatory PCR and qPCR compared to baseline and 3 week supplementation values

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Boston, Massachusetts, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4141001&StudyName=Fecal%20recovery%20of%20the%20probiotic%20bacteria%20Lactobacillus%20rhamnosus%20GG%20%28LGG%29%20and%20Bifidobacterium%20Animalis%20subspecies%20Lactis%20BB-12%20%28BB-12%29